CLINICAL TRIAL: NCT01054742
Title: PREDICT (Part 2)- Prospective Observational Study Of A Cohort Of Naïve Patients With Chronic Hepatitis C Infected With HCV Genotype 1 Low Viral Load (HCV LVL 1) And Treated With Peg-Intron 1.5 ug/Kg/Week Plus Rebetol 800-1200 mg/Day Who Achieved A Negative HCV-RNA At Week 4 and at Week 24
Brief Title: Observational Study of Patients With Chronic Hepatitis C Virus (HCV) Infected With HCV Genotype 1 Low Virus Load (LVL 1) and Effect of PegIntron Plus Rebetol Treatment (Study P04793 Part 2)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04793 Part 2
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood sample for polymerase chain reaction (PCR) Assay
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard of Care PegIntron Plus Ribavirin [Part 2]: Participants who had relapsed during Part 1 of the study, had detectable HCV-RNA on Day 1 of Part 2 of the study, and who were re-treated during Part 2 of the study with standard of care PegIntron plus ribavirin for 48 weeks.
  Interventions: Drug: Standard of Care PegIntron; Drug: Standard of Care Ribavirin

INTERVENTIONS:
Drug: Standard of Care PegIntron — Commercially available PegIntron administered subcutaneously (SC) at 1.5 μg/kg weekly in accordance with the PegIntron Summary of Product Characteristics (SmPC).
  Other Names: peginterferon alfa-2b; PEG2b; SCH 054031
Drug: Standard of Care Ribavirin — Commercially available ribavirin administered orally at 800-1200 mg/day based on body weight in accordance with the ribavirin SmPC.
  Other Names: REBETOL;; SCH 018908

SUMMARY:
The purpose of this observational study was to provide summary data from participants who relapsed at the end of the follow-up phase after 24 weeks of treatment with standard care PegIntron plus ribavirin in Part 1 of the study (NCT00709228) and who then received retreatment during Part 2 of the study. Relapse was defined as having a positive virology result at the Week 24 post-treatment follow-up, after a negative result at the Week 24 end-of-treatment time point. Hepatitis C Virus Ribonucleic Acid (HCV-RNA) levels were measured at Day 1 and Weeks 12, 24, and 48 of the extension, and at Follow-up Week 24.

DETAILED DESCRIPTION:
All study activities were consistent with the EU Directive 2001/20/EC section for non-interventional studies (i.e. observational studies). Medicinal products are prescribed in the usual manner in accordance with the terms of the marketing authorization. The assignment of the participant to a particular therapeutic strategy is not decided in advance by the trial protocol but falls within current practice and the prescription of the medicine is clearly separated from the decision to include the patient in the study.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* 18 years or older, either gender, any race
* Participant has relapsed at the end of the Part 1 follow-up phase (defined as having a positive virology result at 24 weeks of follow-up post treatment after a negative result at the Week 24 end-of-treatment time point)
* Participant considered suitable for treatment per local label
* Investigator considers suitable and participant consents to be treated

Exclusion Criteria:

* Pregnant women or those who plan to become pregnant or sexual partners of women who plan to become pregnant
* Participant does not qualify based on contra-indication, special warning, special population, and/or pregnancy & lactation section of the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only participants who were originally treated in study P04793 and relapsed during the 24 week follow up phase were offered the chance to receive retreatment with PegIntron and ribavirin for up to an additional 48 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants who had relapsed at Follow-up Week 24 of study Part 1, and were enrolled in Part 2 to complete 48 weeks of retreatment.
Groups:
- Standard of Care PegIntron Plus Ribavirin [Part 2]: Participants who had relapsed during Part 1 of the study, had detectable HCV-RNA on Day 1 of Part 2 of the study, and who were re-treated during Part 2 of the study with standard of care PegIntron plus ribivirin for 48 weeks.
Period: Overall Study
Arm/Group | Standard of Care PegIntron Plus Ribavirin [Part 2]
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Standard of Care PegIntron Plus Ribavirin [Part 2]
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  Russian Federation | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable Hepatitis C Virus Ribonucleic Acid (HCV-RNA) Levels During Part 2 of the Study
Description: A quantitative polymerase chain reaction (PCR) assay was used to measure HCV-RNA.
Time Frame: From Day 1, Week 1 [Part 2 ] through Follow-up Week 24 [ Part 2]
Population: Participants who had relapsed during Part 1 of the study, had detectable HCV-RNA on Day 1, Part 2 of the study, and who consented to retreatment.
Measure: Number; unit: participants
Arm/Group | Standard of Care PegIntron Plus Ribavirin [Part 2]
Number analyzed (Participants) | 2
participants
  Day 1, Study Part 2 | 0
  Treatment Week 12, Study Part 2 | 2
  Treatment Week 24, Study Part 2 | 2
  Treatment Week 48, Study Part 2 | 2
  Follow-up Week 24, Study Part 2 | 2

ADVERSE EVENTS:
Arm/Group | Standard of Care PegIntron Plus Ribavirin [Part 2]
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care PegIntron Plus Ribavirin [Part 2] (N=2)
Depression (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to provide forty-five (45) days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication (including, without limitation, slides and text of oral or other public presentations and text of any transmission through any electronic media), which report any results of the Study. The sponsor shall have the right to review and comment on any presentation including editorial rights.